CLINICAL TRIAL: NCT05009888
Title: COVID-19 SARS-CoV-2 Antibody Testing Study
Acronym: SATS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 302225
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other

GROUPS / COHORTS (1):
- Adult KCL IoPPN Staff: Freely consenting Adult KCL Staff attending King's College London, IoPPN, Denmark Hill site will all have an antibody test on finger prick blood. The antibody test will give a rapid result for the presence of IgG or IgM antibodies to COVID-19

SUMMARY:
SATS is a single site feasibility study to assess the practical and psychological feasibility of using rapid COVID antibody testing of blood obtained from fingertip pin-pricks.

DETAILED DESCRIPTION:
SATS is a feasibility study conducted at a single site - King's College London and South London and Maudsley staff working at the Institute of Psychiatry, Psychology and Neuroscience (IoPPN) at Denmark Hill, London, England. The practical and psychological feasibility of using rapid COVID antibody testing of blood obtained from fingertip pin-pricks will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* King's College Staff member
* Aged 18 years or over
* Able to freely give informed consent

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* known to have an infectious disease including a current SARS-CoV-2 infection.
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the research study, or may influence the result of the research study, or the participant's ability to participate in the research study. Examples of disorders or diseases which would be excluded include:

  * Medically diagnosed bleeding disorder;
  * Medically diagnosed platelet disorder;
  * Anticoagulant medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff members based at the Institute of Psychiatry, Psychology and Neuroscience (IoPPN).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Acceptability of performing antibody testing procedures involving a capillary blood sample collected via finger-prick | 1 Year
  o Acceptability would be represented by the number of participants who consent to and complete the antibody testing procedure.
Test validity of the antibody tests that are performed | 1 Year
  the number of completed tests that are valid with a positive/negative IgG/IgM result and confirmed with a positive control line compared with invalid test results as confirmed with a negative control result.

SECONDARY OUTCOMES:
o Representativeness of participants psychological and behavioural reaction to the testing procedure, their test results, and their willingness to be re-tested. | 1 Year
  Assessed by psychometric testing using visual analogue scales
o Representativeness of participants sampled | 1 Year
  This would be assessed using demographic data collected from participant